CLINICAL TRIAL: NCT05965388
Title: Predictive Value of HBV pgRNA on Long-term Outcomes in Hepatitis B Patients Treated With Antiviral Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Wen-hong Zhang (Other)
Collaborators: Shandong Provincial Hospital (Other Government); First Affiliated Hospital Xi'an Jiaotong University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); The Third People's Hospital of Taiyuan (Other); The First People's Hospital of Yunnan (Other); The First Affiliated Hospital of Anhui Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor-Investigator, Wen-hong Zhang, Director of Division ofInfectious Diseases Affiliation: Huashan Hospital, Huashan Hospital
Organization: Huashan Hospital (Other)
Other Study IDs: COMPASS by REASON
Record Dates: First submitted 2023-06-28; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: HBV; HCC
MeSH Terms: interventions — Interferons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collect the serum samples of CHB patients receiving antiviral therapy during long-term follow-up, and detect the concentration of HBV pgRNA in the samples
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic hepatitis B patients treated with nucleoside analogues or interferon: Chronic hepatitis B patients treated with nucleoside analogues or interferon
  Interventions: Drug: nucleoside analogues or interferon

INTERVENTIONS:
Drug: nucleoside analogues or interferon — ETV、TDF、TAF、TAF、IFN-a-2b

SUMMARY:
The goal of this prospective, exploratory, non-intervention, multi-center, real-world study is to investigate the predictive value of HBV pgRNA in the occurrence of long-term outcomes under antiviral therapy in patients with chronic hepatitis B.

Participants will take the necessary clinical examination and blood draw during the patient's treatment and follow-up, and all the treatment is determined by clinicians.

DETAILED DESCRIPTION:
This study is a prospective, exploratory, multi-center, real-world study, with Huashan Hospital as the leading unit. The study includes patients with chronic hepatitis B who have been determined by clinicians to start, or have already taken the first-line treatment { including pegylated interferon [IFN] monotherapy, a potent nucleos(t)ide analogue [NA] monotherapy, two different potent NAs combination therapy, or NA plus IFN combination therapy. The study only collects clinical data and serum samples, without imposing any additional intervention measures or affecting any relevant clinical decisions. The clinical data is collected from the patient's clinical follow-up examination data, without additional visits and auxiliary examinations. Sample collection During the necessary clinical examination and blood draw during the patient's treatment and follow-up, one additional serum separation tube (3ml) was drawn, without additional invasive examination for the patient. The study will follow up with patients for 5 years to explore the relationship between the serum HBV pgRNA level and the endpoint event at different time points.

ELIGIBILITY:
Inclusion Criteria:

* CHB defined as positive hepatitis B surface antigen at least 6 months, or HBV-related histological changes within 1 year if HBsAg positive less than 6 months;
* Age between 18-80 years, gender is not limited；
* Patients with chronic hepatitis B who have been determined by clinicians to start, or have already taken the first-line treatment {including pegylated interferon [IFN] monotherapy, a potent nucleos(t)ide analogue [NA] monotherapy, two different potent NAs combination therapy, or NA plus IFN combination therapy;
* Patient who reads and signs informed consent.

Exclusion Criteria:

* Patients with malignancies other than hepatocellular carcinoma.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B who have been determined by clinicians to start, or have already taken the first-line treatment {including pegylated interferon [IFN] monotherapy, a potent nucleos(t)ide analogue [NA] monotherapy, two different potent NAs combination therapy, or NA plus IFN combination therapy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Diagnosis of hepatocellular carcinoma during the observation period | 5 years
  Number of Participants with Diagnosis of hepatocellular carcinoma

SECONDARY OUTCOMES:
Number of Participants with Diagnosis of participants with decompensation cirrhosis during the observation period | Week 4, Week 12, Week24, Week36, Week48, Week72, Week96, Week120, Week144, Week168, Week192, Week216 and Week240
  Number of Participants with Diagnosis of participants with decompensation cirrhosis
Number of Participants with Diagnosis of participants with liver transplantation during the observation period | Week 4, Week 12, Week24, Week36, Week48, Week72, Week96, Week120, Week144, Week168, Week192, Week216 and Week240
  Number of Participants with Diagnosis of participants with liver transplantation
Number of Participants with Diagnosis of participants with fibrosis regression and progression during the observation period | Week 4, Week 12, Week24, Week36, Week48, Week72, Week96, Week120, Week144, Week168, Week192, Week216 and Week240
  Number of Participants with Diagnosis of participants with fibrosis regression and progression
Number of Participants with Diagnosis of participants with serological response during the observation period | Week 4, Week 12, Week24, Week36, Week48, Week72, Week96, Week120, Week144, Week168, Week192, Week216 and Week240
  Hepatitis B s Antigen (HBsAg) Loss, seroconversion to HBsAg, Hepatitis B s Antigen (HBeAg) Loss (only patients who are HBeAg positive at baseline), and seroconversion to HBeAg

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - the Affiliated Hosptial of Xuzhou Medical University, Xuzhou, Jiangsu
  - Shandong Provincial Hospital of Shandong University, Jinan, Shandong
  - The Third People's Hospital of Taiyuan, Taiyuan, Shanxi
  - First Affiliated Hospital Xi'an Jiaotong University, Xi’an, Shanxi
  - The First People's Hospital Of YunNan, Kunming, Yunnan
  - Huashan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schweitzer A, Horn J, Mikolajczyk RT, Krause G, Ott JJ. Estimations of worldwide prevalence of chronic hepatitis B virus infection: a systematic review of data published between 1965 and 2013. Lancet. 2015 Oct 17;386(10003):1546-55. doi: 10.1016/S0140-6736(15)61412-X. Epub 2015 Jul 28. PMID 26231459
- [Background] Chinese Society of Infectious Diseases, Chinese Medical Association; Chinese Society of Hepatology, Chinese Medical Association. [The guidelines of prevention and treatment for chronic hepatitis B (2019 version)]. Zhonghua Gan Zang Bing Za Zhi. 2019 Dec 20;27(12):938-961. doi: 10.3760/cma.j.issn.1007-3418.2019.12.007. Chinese. PMID 31941257
- [Background] Jung MC, Pape GR. Immunology of hepatitis B infection. Lancet Infect Dis. 2002 Jan;2(1):43-50. doi: 10.1016/s1473-3099(01)00172-4. PMID 11892495
- [Background] Shin EC, Sung PS, Park SH. Immune responses and immunopathology in acute and chronic viral hepatitis. Nat Rev Immunol. 2016 Aug;16(8):509-23. doi: 10.1038/nri.2016.69. Epub 2016 Jul 4. PMID 27374637
- [Background] Nassal M. HBV cccDNA: viral persistence reservoir and key obstacle for a cure of chronic hepatitis B. Gut. 2015 Dec;64(12):1972-84. doi: 10.1136/gutjnl-2015-309809. Epub 2015 Jun 5. PMID 26048673
- [Background] Pollicino T, Belloni L, Raffa G, Pediconi N, Squadrito G, Raimondo G, Levrero M. Hepatitis B virus replication is regulated by the acetylation status of hepatitis B virus cccDNA-bound H3 and H4 histones. Gastroenterology. 2006 Mar;130(3):823-37. doi: 10.1053/j.gastro.2006.01.001. PMID 16530522
- [Background] Ko C, Chakraborty A, Chou WM, Hasreiter J, Wettengel JM, Stadler D, Bester R, Asen T, Zhang K, Wisskirchen K, McKeating JA, Ryu WS, Protzer U. Hepatitis B virus genome recycling and de novo secondary infection events maintain stable cccDNA levels. J Hepatol. 2018 Dec;69(6):1231-1241. doi: 10.1016/j.jhep.2018.08.012. Epub 2018 Aug 22. PMID 30142426
- [Background] Tang LSY, Covert E, Wilson E, Kottilil S. Chronic Hepatitis B Infection: A Review. JAMA. 2018 May 1;319(17):1802-1813. doi: 10.1001/jama.2018.3795. PMID 29715359
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] Omata M, Cheng AL, Kokudo N, Kudo M, Lee JM, Jia J, Tateishi R, Han KH, Chawla YK, Shiina S, Jafri W, Payawal DA, Ohki T, Ogasawara S, Chen PJ, Lesmana CRA, Lesmana LA, Gani RA, Obi S, Dokmeci AK, Sarin SK. Asia-Pacific clinical practice guidelines on the management of hepatocellular carcinoma: a 2017 update. Hepatol Int. 2017 Jul;11(4):317-370. doi: 10.1007/s12072-017-9799-9. Epub 2017 Jun 15. PMID 28620797
- [Background] Kim GA, Lim YS, An J, Lee D, Shim JH, Kim KM, Lee HC, Chung YH, Lee YS, Suh DJ. HBsAg seroclearance after nucleoside analogue therapy in patients with chronic hepatitis B: clinical outcomes and durability. Gut. 2014 Aug;63(8):1325-32. doi: 10.1136/gutjnl-2013-305517. Epub 2013 Oct 25. PMID 24162593
- [Background] Lim TH, Gane E, Moyes C, Borman B, Cunningham C. HBsAg loss in a New Zealand community study with 28-year follow-up: rates, predictors and long-term outcomes. Hepatol Int. 2016 Sep;10(5):829-37. doi: 10.1007/s12072-016-9709-6. Epub 2016 Mar 8. PMID 26957439
- [Background] Wang YX, Niklasch M, Liu T, Wang Y, Shi B, Yuan W, Baumert TF, Yuan Z, Tong S, Nassal M, Wen YM. Interferon-inducible MX2 is a host restriction factor of hepatitis B virus replication. J Hepatol. 2020 May;72(5):865-876. doi: 10.1016/j.jhep.2019.12.009. Epub 2019 Dec 18. PMID 31863794
- [Background] Tan G, Yi Z, Song H, Xu F, Li F, Aliyari R, Zhang H, Du P, Ding Y, Niu J, Wang X, Su L, Qin FX, Cheng G. Type-I-IFN-Stimulated Gene TRIM5gamma Inhibits HBV Replication by Promoting HBx Degradation. Cell Rep. 2019 Dec 10;29(11):3551-3563.e3. doi: 10.1016/j.celrep.2019.11.041. PMID 31825835
- [Background] Sadler AJ, Williams BR. Interferon-inducible antiviral effectors. Nat Rev Immunol. 2008 Jul;8(7):559-68. doi: 10.1038/nri2314. PMID 18575461
- [Background] Marcellin P, Ahn SH, Ma X, Caruntu FA, Tak WY, Elkashab M, Chuang WL, Lim SG, Tabak F, Mehta R, Petersen J, Foster GR, Lou L, Martins EB, Dinh P, Lin L, Corsa A, Charuworn P, Subramanian GM, Reiser H, Reesink HW, Fung S, Strasser SI, Trinh H, Buti M, Gaeta GB, Hui AJ, Papatheodoridis G, Flisiak R, Chan HL; Study 149 Investigators. Combination of Tenofovir Disoproxil Fumarate and Peginterferon alpha-2a Increases Loss of Hepatitis B Surface Antigen in Patients With Chronic Hepatitis B. Gastroenterology. 2016 Jan;150(1):134-144.e10. doi: 10.1053/j.gastro.2015.09.043. Epub 2015 Oct 8. PMID 26453773
- [Background] Reijnders JG, Rijckborst V, Sonneveld MJ, Scherbeijn SM, Boucher CA, Hansen BE, Janssen HL. Kinetics of hepatitis B surface antigen differ between treatment with peginterferon and entecavir. J Hepatol. 2011 Mar;54(3):449-54. doi: 10.1016/j.jhep.2010.07.046. Epub 2010 Nov 5. PMID 21112655
- [Background] Wursthorn K, Lutgehetmann M, Dandri M, Volz T, Buggisch P, Zollner B, Longerich T, Schirmacher P, Metzler F, Zankel M, Fischer C, Currie G, Brosgart C, Petersen J. Peginterferon alpha-2b plus adefovir induce strong cccDNA decline and HBsAg reduction in patients with chronic hepatitis B. Hepatology. 2006 Sep;44(3):675-84. doi: 10.1002/hep.21282. PMID 16941693
- [Background] van Bommel F, van Bommel A, Krauel A, Wat C, Pavlovic V, Yang L, Deichsel D, Berg T, Bohm S. Serum HBV RNA as a Predictor of Peginterferon Alfa-2a Response in Patients With HBeAg-Positive Chronic Hepatitis B. J Infect Dis. 2018 Aug 24;218(7):1066-1074. doi: 10.1093/infdis/jiy270. PMID 29741634
- [Background] Huang YW, Takahashi S, Tsuge M, Chen CL, Wang TC, Abe H, Hu JT, Chen DS, Yang SS, Chayama K, Kao JH. On-treatment low serum HBV RNA level predicts initial virological response in chronic hepatitis B patients receiving nucleoside analogue therapy. Antivir Ther. 2015;20(4):369-75. doi: 10.3851/IMP2777. Epub 2014 Apr 16. PMID 24739420
- [Background] Jansen L, Kootstra NA, van Dort KA, Takkenberg RB, Reesink HW, Zaaijer HL. Hepatitis B Virus Pregenomic RNA Is Present in Virions in Plasma and Is Associated With a Response to Pegylated Interferon Alfa-2a and Nucleos(t)ide Analogues. J Infect Dis. 2016 Jan 15;213(2):224-32. doi: 10.1093/infdis/jiv397. Epub 2015 Jul 27. PMID 26216905
- [Background] Tsuge M, Murakami E, Imamura M, Abe H, Miki D, Hiraga N, Takahashi S, Ochi H, Nelson Hayes C, Ginba H, Matsuyama K, Kawakami H, Chayama K. Serum HBV RNA and HBeAg are useful markers for the safe discontinuation of nucleotide analogue treatments in chronic hepatitis B patients. J Gastroenterol. 2013 Oct;48(10):1188-204. doi: 10.1007/s00535-012-0737-2. Epub 2013 Feb 9. PMID 23397114
- [Background] Serum hepatitis B virus RNA levels as an early predictor of hepatitis B envelope antigen seroconversion during treatment with polymerase inhibitors. Hepatology. 2016 Jan;63(1):349. doi: 10.1002/hep.28349. No abstract available. PMID 26689731
- [Background] Department of Medical Administration, National Health and Health Commission of the People's Republic of China. [Guidelines for diagnosis and treatment of primary liver cancer in China (2019 edition)]. Zhonghua Gan Zang Bing Za Zhi. 2020 Feb 20;28(2):112-128. doi: 10.3760/cma.j.issn.1007-3418.2020.02.004. No abstract available. Chinese. PMID 32164061
- [Background] Chinese Society of Hepatology,Chinese Medical Association. [Chinese guidelines on the management of liver cirrhosis]. Zhonghua Gan Zang Bing Za Zhi. 2019 Nov 20;27(11):846-865. doi: 10.3760/cma.j.issn.1007-3418.2019.11.008. Chinese. PMID 31941240